CLINICAL TRIAL: NCT06132347
Title: Performances of DendrisCHIP®OA in Bone and Joint Infections
Acronym: DENDRIS
Status: Withdrawn | Type: Observational
Why Stopped: The company that supplies the Medical Device has withdrawn.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: ARX-DENDRIS
Record Dates: First submitted 2023-10-27; First posted 2023-11-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Bone Infection; Joint Infection; Molecular Diagnostic
Keywords: Bone and joint infection; Molecular diagnostic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bone and joint infections (BJI) with and without prosthetic material (knee, hip and shoulder) are complex to diagnose and treat, justifying the creation of expert centers by the French Ministry of Health (CRIOAc).

In case of BJI with material, the diagnosis is based on a set of clinical, bacteriological, cytological and radiological criteria known as the EBJIS 2021 (European Bone & Joint Infections Society) criteria. For septic arthritis, diagnosis is based on bacteriology and cytology.

Microbiology remains essential, and the delay of obtention of microbiological results is crucial to adapt the antibiotic treatment. Although, culture-based microbiology remains the most common diagnosis of BJI, its regular failure to identify the causative pathogen as well as its long-term modus operandi motivates the development of rapid and accurate molecular methods.

The DendrisCHIP®OA platform has demonstrated its ability to offer routine molecular identification of the current micro-organisms involved in BJI, in less than 5 hours, with the detection of mecA resistance genes on series of 16 to 64 samples . The DendrisCHIP®OA is CE-marked and has already been the subject of an initial publication evaluating its performance in a single center.

The main objective of this study is to evaluate the diagnostic performances of the DendrisCHIP®OA in detecting the pathogens recognized in its panel and the detection of the mecA gene compared with the routine microbiological techniques used in the inclusion centers participating to the study.

The study aims to include 100 patients during 6 months in five inclusion centers in the Ile de France region.

DETAILED DESCRIPTION:
Bone and joint infections (BJI) with and without prosthetic material (knee, hip and shoulder) are complex to diagnose and treat, justifying the creation of expert centers by the French Ministry of Health (CRIOAc).

In case of BJI with material, the diagnosis is based on a set of clinical, bacteriological, cytological and radiological criteria known as the EBJIS 2021 (European Bone & Joint Infections Society) criteria. For septic arthritis, diagnosis is based on bacteriology and cytology.

Currently, a patient with suspected BJI remains hospitalized for at least 5 days with parenteral antibiotics, until the results of bacteriological culture. If the bacteriological diagnosis is negative, and the clinical suspicion of infection is weak, treatment is stopped at least 7 days post-operatively. If the microbiological diagnosis is positive, the choice of the therapeutic will depend on the isolated bacterial species. So, microbiology remains essential, and the delay of obtention of microbiological results is crucial to adapt the antibiotic treatment.

Microbiological culture techniques remain the gold standard, but are time-consuming (3 to 14 days), and require qualified personnel, with a risk of false negative results in 5 to 10% of cases (prior antibiotic therapy, atypical or fastidious microorganisms). These diagnostic limitations lead to care difficulties, with major consequences in terms of morbidity, quality of life and treatment costs.

Syndromic molecular methods (metagenomics, Unyvero Cartridges, Biofire® nested-PCR), which could improve microbiological diagnosis, are currently being evaluated, but have a number of drawbacks that make this tests as complementary methods in specialized laboratories (cost, productivity, insufficient panels, etc.).

The DendrisCHIP®OA platform has demonstrated its ability to offer routine molecular identification of the current micro-organisms involved in BJI, in less than 5 hours, with the detection of mecA resistance genes on series of 16 to 64 samples. The DendrisCHIP®OA is CE-marked and has already been the subject of an initial publication evaluating its performances in a single center.

On the other hand, the innovation brought by this technology is the analysis by artificial intelligence thanks to the DendriSOFT software, which takes into account biological variability. This database is constantly enhanced by self-learning.

The research will be carried out over a 6-months period to include 100 patients in five inclusion centers (CRIOAc) in Ile de France region, with a minimum of 2 patients treated for BJI per week per inclusion center.

The main objective of this study is to evaluate the diagnostic performances of the DendrisCHIP®OA in detecting the pathogens recognized in its panel and the detection of the mecA gene compared with the routine microbiological techniques used in the inclusion centers participating to the study.

The secondary objectives are :

* to document discrepancies using alternative techniques (specific PCR, sequencing)
* to compare turnaround times (from sampling to biological validation) between the routine microbiological technique and DendrisCHIP®OA
* to evaluate the impact on the patient's therapeutic management (modification of antibiotic treatment)
* to evaluate diagnostic performance of the DendrisCHIP®OA on a sub-group of culture-negative patients with clinical signs of infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ⩾ 18 years,
* Patients suspected of bone and joint infection,
* Any patient who had intraoperative samples for suspected BJI with or without material, and who received on broad-spectrum antibiotic therapy post-operatively,
* No opposition from the patient, or its surrounding.

Exclusion Criteria:

* Refusal to participate,
* Pregnant or beastfeeding,
* Patient under guardianship or curatorship,
* Patient not affiliated to social security,
* Patient affiliated to the Aide Médicale d'Etat (AME).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had intraoperative samples for suspected BJI with or without material, and who received on broad-spectrum antibiotic therapy post-operatively.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performances | at 6 months
  Diagnostic performance of the DendrisCHIP®OA OA method in routine situation compared with the laboratory's usual method according to method validation criteria (sensitivity, specificity, NPV, PPV).

SECONDARY OUTCOMES:
Document discrepancies using alternative techniques (specific PCR, sequencing) | through study completion, an average of 6 months
  Document discrepancies, in case of discrepancy between the DendrisCHIP®OA test result and the reference microbiological method.
  The frozen sample is process for additional techniques (specific PCR or universal 16S PCR with sequencing).
Difference of delay | at 6 months
  Comparing of the delay between sampling date and date of biological validation, of DendrisCHIP®OA test and routine microbiological method.
Impact evaluation of antibiotic therapy | at 6 months
  Duration of parenteral antibiotic therapy and time to adapt antibiotic treatment to microbiological documentation.
Performance evaluation on a subgroup | at the end of study, in an average of 6 months
  Determination of the sensitivity, specificity, PPV and NPV of the DendrisCHIP®OA method on a subgroup of patients negative with the routine microbiological technique but with clinical signs of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Roux, PharmD, PhD, Principal Investigator — Laboratory of microbiology, Ambroise Paré hospital - APHP